CLINICAL TRIAL: NCT06362486
Title: Stress in Pregnancy During the Covid19 Pandemic and Impact on the Newborn Neurodevelopment
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: SIGNATURE
Record Dates: First submitted 2024-04-11; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-02

CONDITIONS: Covid19 and Pregnancy
MeSH Terms: conditions — COVID-19 | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — A group of newborns of mothers infected by sars-cov-2 will present biological markers suggestive of presenting an abnormal inflammatory state (inflammation signature) that puts them at risk of suffering neurodevelopmental alterations. Inflammatory alterations in NBs will be related to clinical variables such as the time (gestational age) of maternal infection and its severity and, based on previous literature, alterations in the innate immune response will be associated with the clinical phenotype of the newborn. This is the cohort C N=100 (infected and non-infected)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A N=1000: neurodevelopment assessment by pediatrician, need to refer to neurodevelopmental assessment by specialized team. m-chat. autism diagnosis.
  Interventions: Other: Severity of infection, time of infection.
- Cohort B N=500: Mental health assessment
  Interventions: Other: Mental health assessment
- Cohort C N=100: biological
  Interventions: Other: biological

INTERVENTIONS:
Other: Severity of infection, time of infection. — Severity of infection, time of infection.
  Groups: Cohort A N=1000
Other: Mental health assessment — Mental health assessment
  Groups: Cohort B N=500
Other: biological — Prognostic immunologic factors associated with cognitive impairment in children born of sars-cov-2-infected mothers.
  Groups: Cohort C N=100

SUMMARY:
The Covid19 pandemic, paradoxically, represents a valuable opportunity to carry out cohort studies that allow us to advance our knowledge about the relationship between inflammation, brain development and an increased risk of suffering from neuropsychiatric disorders or alterations. In addition, the current availability of sophisticated biological techniques and evaluation procedures represents an unique option for this purpose.

Here, we propose a cohort study of sars-cov-2 (type 2 coronavirus causing severe acute respiratory syndrome) infected pregnant women and newborns. We will try to answer the following questions: (i) what is the inflammatory / immune status of newborns (NBs) of mothers infected by Covid19 like?; (ii) is there a relationship between the clinical characteristics of the maternal infection (severity / moment / of infection) and the inflammatory status of the newborn?; (iii) could these features increase the vulnerability to developing central nervous system (CNS) alterations at an early age, and at some point during adult life ?; (iv) How is the Covid19 infected mother's placenta altered? Do the placental alterations Covid19 mediated contribute to develop CNS alterations?; (v) is the infection associated with phenotypes obtained through neurological and neurodevelopmental clinical evaluation (hypotonia, clumsiness, impaired communication and sociability) in children at 6 months and 12 months?

Our main objective is to explore how the presence of stressors and prenatal sars-cov-2 infection generates an abnormal inflammatory activity in the newborn, which is associated with neurodevelopmental disorders and which confers a greater risk of developing neuropsychiatric disorders. The biological information of the umbilical cord (fetus blood) and peripheral blood of the mother obtained after childbirth was provided by the cohort of women during the Covid19 pandemic monitored during their pregnancy, delivery, childbirth and postpartum. These samples and the clinical characterisation of the cohort of mothers and newborns, of which we will be able to do an exhaustive longitudinal follow-up, are tremendously valuable at this time. There is a need to establish new research strategies to understand the pathophysiology of neuropsychiatric diseases, and to discover new molecular and cellular mechanisms involved in the development of the CNS.

ELIGIBILITY:
Inclusion Criteria:

* 1. over 18 years old
* 2. Ultrasound-confirmed pregnancy
* 3. infected (past or present) or non-infected with Covid19

Exclusion Criteria:

* 1. presents alcohol abuse during pregnancy
* 2. other concomitant causes of risk of demonstrated neurodevelopmental disorders
* 3. presents drug abuse except tobacco during pregnancy
* 4. under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women over 18 years of age, without concomitant diseases that affect the neurodevelopment of the newborn or use of toxic substances. For the data collection of the CASE group, these women must have been or be positive for Covid-19. For the CONTROL group, the pregnant woman must not have been infected by Covid-19.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
explore how the presence of stressors and prenatal sars-cov-2 infection generates an abnormal inflammatory activity in the newborn | birth, at 6 months and 12 months
  explore how the presence of stressors and prenatal sars-cov-2 infection generates an abnormal inflammatory activity in the newborn, which is associated with neurodevelopmental disorders and which confers a greater risk of developing neuropsychiatric disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain